CLINICAL TRIAL: NCT02623413
Title: Cohort Study of German Hematological / Oncological Wards to Assess the Effect of Contact Precautions on Nosocomial Colonization With Vancomycin Resistant Enterococci
Acronym: CONTROL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Cologne (Other)
Collaborators: German Center for Infection Research (Other); University Hospital Tuebingen (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Freiburg (Other); Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Maria J.G.T. Vehreschild, PD Dr., University of Cologne
Other Study IDs: CONTROL
Record Dates: First submitted 2015-11-23; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Vancomycin (Glycopeptide) Resistant Enterococcus (VRE); Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cultured VRE strains from rectal swabs, stool samples and infection sites.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sites implementing contact precautions: Centers isolating for VRE may only participate if complying with the following standards:
  * Contact precautions triggered by the initial detection of VRE
  * Patients discharged as a VRE-carrier must be placed in contact isolation upon readmission
  * Termination of contact precautions after at least two consecutive VRE-negative consecutive fecal screening cultures
  * Resumption of contact isolation on first subsequent VRE-positive culture
  Contact precautions must encompass the following measures:
  * Patients: Placement in single rooms. Cohorting is only permitted, in case of unavailability of single rooms
  * Staff and visitors: Wearing of gloves and gowns when entering the room.
  * Patients: Wearing of gloves and gowns when leaving the room.
- Sites not implementing contact precautions: Only VRE colonized or infected patients with urinary or fecal incontinence or diarrhea (defined as > 3 loose bowel movements/day), must be isolated in single rooms at any time during the study.

SUMMARY:
The study aims to evaluate the impact of contact precautions on the rate of VRE- the rate of colonization and infection aand hospital-acquired VRE transmissions.

Hematological and oncological wards in hospitals with a non-outbreak setting for VRE and adhering to at least the following standard of care are eligible for study participation:

Fecal screening for the presence of VRE of all patients within 72 hours of each admission by use of a rectal swab or stool sample Follow-up fecal screening once a week and within 72 hours of discharge Implementation of clinical standards aimed at VRE decolonization is not allowed on wards participating in this study, including in the context of clinical studies.

Sites will be grouped according to their approach regarding contact isolation (see group description).

As a control for external factors a hand hygiene program, including training and adherence assessments, will be implemented.

This observational study prospectively compares wards with different approaches to isolation. All screening and isolation measures are already in place on participating wards (i.e. constituted a site selection criterion) and are exclusively implemented as part of the standard of care. Sites are free to adjust their standard of care as they see fit. No intervention will be performed.

ELIGIBILITY:
* Inclusion criteria:

  * Inpatient hospitalization during the study period on one of the participating wards.
* Exclusion criteria:

  * None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated on one of the participating wards
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital-acquired VRE-colonization and/or infection | 1 year

SECONDARY OUTCOMES:
Incidence of patient-to-patient transmission of VRE | 1 year
  Defined by the isolation of molecularly related VRE strains from patients with overlapping hospitalization periods in the same ward.
Incidence of VRE intestinal colonization among all patients | 1 year
  Colonization is defined as the isolation of VRE from fecal screening samples
Incidence of VRE bloodstream infections among all patients | 1 year
  VRE bloodstream infection is defined by the isolation of VRE from at least one blood culture
Incidence of VRE bloodstream infections among previously colonized patients | 1 year
Readmission fraction associated with VRE infection | 1 year
Prevalence of VRE in the community. | 1 year
  Defined as VRE-colonization upon the first admission of a patient not transferred from another hospital or a long term care facility